CLINICAL TRIAL: NCT02101905
Title: Drug Distribution and Pharmacodynamic Study of Pulsatile Lapatinib in Surgically Accessible EGFR-Amplified Recurrent High-Grade Glioma
Brief Title: Lapatinib Ditosylate Before Surgery in Treating Patients With Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00634; NCI-2014-00634 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ABTC-1302 (Other: Adult Brain Tumor Consortium); ABTC-1302 (Other: CTEP); U01CA137443 (NIH); UM1CA137443 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Ependymoma; Anaplastic Oligodendroglioma; Gliosarcoma; Mixed Glioma; Recurrent Adult Brain Neoplasm; Recurrent Glioblastoma
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Gliosarcoma; Glioma; Brain Neoplasms; Glioblastoma | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (lapatinib ditosylate, surgery) (Experimental): Patients receive lapatinib ditosylate PO BID on days -2 to 0. Within 3-5 hours after last dose of lapatinib ditosylate, patients undergo surgical resection of tumor on day 0. Within 30 days of surgical resection of tumor, patients receive lapatinib ditosylate BID for 2 days every 7 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lapatinib; Drug: Lapatinib Ditosylate; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery
- Reference Group (surgery, lapatinib ditosylate) (Active Comparator): Patients undergo surgery on day 0. Within 30 days of surgical resection of tumor, patients receive lapatinib ditosylate BID for 2 days every 7 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lapatinib; Drug: Lapatinib Ditosylate; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lapatinib — Given PO
  Other Names: GSK572016; GW 2016; GW 572016; GW-572016; GW2016; GW572016
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
Other: Pharmacological Study — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection of tumor

SUMMARY:
This pilot phase I clinical trial studies how well lapatinib ditosylate before surgery works in treating patients with high-grade glioma that has come back after a period of time during which the tumor could not be detected. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To achieve an intratumoral lapatinib (lapatinib ditosylate) concentration of at least 1.5 uM in at least 70% of patients 3 hours after the last dose of pulsatile lapatinib. (Group A) II. To determine the pharmacodynamic (PD) effect of pulsatile lapatinib (at pulsatile maximum tolerated dose [MTD]) on epidermal growth factor receptor (EGFR) phosphorylation (using Mesoscale Discovery enzyme-linked immunosorbent assay [ELISA] assay for total and phospho-EGFR). (Group A and Reference Group)

SECONDARY/EXPLORATORY OBJECTIVES:

Ia. To evaluate the safety profile of pulsatile lapatinib in pre-operative patients with EGFR amplified recurrent high-grade glioma. (Group A and Reference Group) Ib. To evaluate acute and late toxicities associated with pulsatile lapatinib. (Group A and Reference Group) II. To determine the effect of lapatinib on tumor cell proliferation (marker of proliferation Ki-67 [KI-67] staining). (Group A compared to Reference Group) III. To determine the ex-vivo sensitivity of tumor sphere cultures to lapatinib. (Group A and Reference Group) IV. To assess tumor objective response rate (ORR). (Group A and Reference Group) V. To estimate overall survival (OS). (Group A and Reference Group) VI. To estimate progression-free survival. (Group A and Reference Group)

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

GROUP A: Patients receive lapatinib ditosylate orally (PO) twice daily (BID) on days -2 to 0. Within 3-5 hours after last dose of lapatinib ditosylate, patients undergo surgical resection of tumor on day 0. Within 30 days of surgical resection of tumor, patients receive lapatinib ditosylate BID for 2 days every 7 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

REFERENCE GROUP: Patients undergo surgical resection of tumor on day 0. Within 30 days of surgical resection of tumor, patients receive lapatinib ditosylate BID for 2 days every 7 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at 30 days, every 2 months for 2 years, and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven World Health Organization (WHO) grade IV glioblastoma/ gliosarcoma or WHO grade III glioma (anaplastic astrocytoma, anaplastic oligodendroglioma, mixed anaplastic oligoastrocytoma, anaplastic ependymoma) which is progressive or recurrent following radiation therapy +/- chemotherapy
* Patients must have measurable, supratentorial contrast-enhancing progressive or recurrent high-grade glioma by magnetic resonance imaging (MRI) imaging within 21 days of starting treatment; patient must be able to tolerate MRIs
* Patients may have an unlimited number of prior therapy regimens
* Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 4 weeks from the last treatment with bevacizumab
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent other than bevacizumab (e.g., hydroxychloroquine, etc.)
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers; patients must be eligible for surgical resection according to the following criteria:

  * Expectation that the surgeon is able to resect at least 500 mg of tumor from enhancing tumor and 100 mg from non-enhancing tumor with low risk of inducing neurological injury
* Patient tumor sample must have evidence of EGFR gene amplification by fluorescence in situ hybridization (FISH) using a Clinical Laboratory Improvement Act (CLIA)-certified laboratory assay
* Paraffin embedded tissue must be available from initial surgical resection at diagnosis (prior to any treatment)
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Activated partial thromboplastin time (APTT)/partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
* Patients must have left ventricular ejection fraction (LVEF) within normal institutional limits within 21 days of starting treatment
* Patients must have a 12-lead electrocardiogram performed within 2 weeks of treatment start with corrected (QTC) =< 470 msec
* Patients must be able to provide written informed consent
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry; women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after completion of lapatinib administration
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
* Patients must be able to swallow medication by mouth, either tablets or dispersed tablets in solution

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib are ineligible
* Patients with prior therapy with EGFR inhibitors are ineligible because treatment with EGFR kinase inhibitors or other EGFR-targeted agents has the potential to deplete the tumor of EGFR-amplified or EGFR mutant cell populations and confound the evaluation of lapatinib effects on EGFR phosphorylation; patients with prior EGFRvIII vaccine are eligible if recurrent tumor is positive for EGFR gene amplification
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol; patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of lapatinib
* Patients must not have evidence of significant hematologic, renal, or hepatic dysfunction
* Patients must not have evidence of significant intracranial hemorrhage
* Patients with uncontrolled intercurrent illness including, but not limited to, hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study because lapatinib has potential for teratogenic or abortifacients effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lapatinib, breastfeeding should be discontinued if the mother is treated with lapatinib
* Human immunodeficiency virus (HIV)-positive patients on strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers or inhibitors are ineligible
* Patients who have acute or currently active/requiring anti-viral therapy hepatic or biliary disease are ineligible (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases from the primary brain tumor, or stable chronic liver disease per investigator assessment)
* Patients receiving P-glycoprotein (P-gp) inhibitors are ineligible
* Patients who are receiving a drug that has a risk of QTc prolongation if QTc is >= 460 msec. are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
To Determine the Lapatinib Ditosylate Intratumoral Concentration (Pharmacokinetics) | Baseline and day of surgery
  4 pk samples obtained: pretreatment, pre-surgery, post-surgery and interpolated pre-surgery each subject received 2500mg twice a day for two days.
To Determine the Ratio of Phosphorylated (p)EGFR/Total EGFR (PD) in Tumor Tissue | Day of surgery
  A ratio of pEGFR/total EGFR at 80% reduction from a median value from the untreated reference group will be considered as the putative threshold to qualify a near complete inhibition of EGFR (at 80%).

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to day 30
  Will be assessed by NCI CTCAE. All Treatment or surgically related AEs will be reported descriptively. A proportion of toxicity equal or greater than 3 will be estimated using binomial distribution.
Inhibition of tumor cell proliferation (KI-67) | Inhibition of Tumor Cell Proliferation (KI-67)
  Descriptive statistics will be used for summarizes results and Box plots could be used to present the difference between the treated and untreated groups.
  This was more an explorative measure and it was not completed.
Ex-vivo Sensitivity of Tumor Sphere Cultures to Lapatinib Ditosylate | Day of surgery
  The ex-vivo sensitivity of tumor sphere cultures established from surgical specimens to pulsatile lapatinib ditosylate is defined by a minimum of 20% reduction in cell proliferation as measured by cell titer glow in the pulsatile lapatinib ditosylate group compared to the untreated group. Fisher's exact test will be used for testing a difference in the proportion between the two groups.
  This was more an explorative measure and it was not completed.
Objective Response Rate | Up to 2 years
  Will be estimated along with 95% confidence intervals using the exact binomial method.
Overall Survival | From the date of treatment start to the date of death, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate overall survival probability and median time of survival along with a 95% confidence interval.
Progression-free Survival | Start of treatment up to 6 months
  The Kaplan-Meier method will be used to estimate progression-free survival probability and median time of survival along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F Cloughesy, Principal Investigator — National Cancer Institute (NCI)
Locations (12):
- United States (12):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02101905/Prot_SAP_000.pdf